CLINICAL TRIAL: NCT05086536
Title: Re-compensation and Its Clinical Characteristics in Treatment-naïve HBV Decompensated Cirrhosis on Antiviral Therapy
Brief Title: Re-compensation and Its Clinical Characteristics in HBV Decompensated Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing YouAn Hospital (Other); Shandong Provincial Hospital (Other Government); The Affiliated Hospital of Qingdao University (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Xiangya Hospital of Central South University (Other); The Second Affiliated Hospital of Baotou Medical College (Other)
Responsible Party: Principal Investigator, Hong You, Vice director, Beijing Friendship Hospital
Other Study IDs: 2021-P2-224-01
Record Dates: First submitted 2021-09-19; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Hepatitis B; Decompensated Cirrhosis
Keywords: re-compensation; treatment-naive; HBV; decompensation
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- early stage decompensation cohort: Patients occurred first decompensated events and initiating nucleoside analogs (NUCs) based treatment within 3 months were retrospectively included.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — This is a retrospective and observational study.

SUMMARY:
In this study, treatment-naïve HBV-related cirrhosis patients were retrospectively enrolled at the first episode of decompensation (ascites or variceal hemorrhage). Patients were followed up every 6 months until death /liver transplantation or for 5 years. Clinical data from medical records about past history, first decompensated events, second /further decompensated events, HCC, and death/ liver transplantation were retrospectively collected. In this retrospective study, the incidence of re-compensation and its clinical characteristics were mainly explored.

DETAILED DESCRIPTION:
In this study, treatment-naïve HBV-related cirrhosis patients were retrospectively enrolled at the first episode of decompensation (ascites or variceal hemorrhage). Patients were followed up every 6 months until death /liver transplantation or for 5 years. WBC, RBC, HGB, PLT, CRP, PT, PTA, INR, ALT, AST, TB, DB, ALB, GLO, ALP, GGT, CHE, BUN, Cr, Na, GLU, CHOL, TG, HDL-C, LDL-C, AFP, HBsAg, HBV-DNA, LSM, BUS, MRI/CT and gastroscope from medical records about past history, first decompensated events, second /further decompensated events, HCC, and death/ liver transplantation were retrospectively collected. This retrospective study aimed to explore the incidence of re-compensation and its clinical characteristics.

ELIGIBILITY:
Inclusion Criteria:

1. Ascites and/or variceal hemorrhage (VH) as the first decompensated events;
2. Initiating antiviral therapy within 3 months of the first decompensated events;
3. Clinical parameters were available at the first decompensated events, including PLT, ALT, ALB, TB, PT/INR, Cr, HBV DNA, BUS,
4. Clinical outcomes were classified:

   1. Without further decompensation: medical records at year-1, year 2 to 4, and year-5 were available.
   2. With ≥ 2 episodes of decompensation: medical records for decompensation were available.

Exclusion Criteria:

1. Hepatocellular carcinoma prior to /within 6 months of first decompensated events;
2. Liver transplantation /death within 6 months of first decompensated events;
3. complicated with other chronic liver diseases, including HCV, DILI, AIH, NAFLD, ALD.
4. Any complication of severe heart, lung, kidney, brain, blood diseases or other severe systematic diseases;
5. Pregnant women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HBV-decompensated cirrhosis patients who occurred first decompensated events and initiated antiviral therapy within 3 months.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-10-15 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of re-compensation | Year 5
  Patients who did not occur further decompensation

SECONDARY OUTCOMES:
Cumulative incidence of re-compensation | Year 1, 2, 3, and 4
  Patients who did not occur further decompensation
Annual incidence of second decompensation | Year 1, 2, 3, 4, and 5
  Patients who occurred second decompensation
Cumulative incidence of liver-related death / liver transplantation | Year 1, 2, 3, 4, and 5
  Patients who died of decompensation
Cumulative incidence of HCC | Year 1, 2, 3, 4, and 5
  Patients who occurred HCC
Dynamic changes of Child-Pugh score in re-compensated and not re-compensated group | Year 1, 2, 3, 4, and 5
  Child-Pugh
Dynamic changes of MELD score in re-compensated and not re-compensated group | Year 1, 2, 3, 4, and 5
  MELD
Dynamic changes of APRI score in re-compensated and not re-compensated group | Year 1, 2, 3, 4, and 5
  APRI
Dynamic changes of FIB-4 score in re-compensated and not re-compensated group | Year 1, 2, 3, 4, and 5
  FIB-4
Dynamic changes of liver stiffness values measured by Transient Elastography in re-compensated and not re-compensated group | Year 1, 2, 3, 4, and 5
  Liver stiffness

CONTACTS AND LOCATIONS:
Overall Officials: Hong You, Doctor, Principal Investigator — Beijing Friendship Hospita
Locations (7):
- China (7):
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing YouAn Hospital, Capital Medical University, Beijing, Beijing Municipality
  - XiangYa Hospital Central South University, Changsha, Hunan
  - The Second Affiliated Hospital of Baotou Medical Coll, Baotou, Inner Mongolia
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jang JW, Choi JY, Kim YS, Woo HY, Choi SK, Lee CH, Kim TY, Sohn JH, Tak WY, Han KH. Long-term effect of antiviral therapy on disease course after decompensation in patients with hepatitis B virus-related cirrhosis. Hepatology. 2015 Jun;61(6):1809-20. doi: 10.1002/hep.27723. Epub 2015 Mar 18. PMID 25627342
- [Background] Belli LS, Berenguer M, Cortesi PA, Strazzabosco M, Rockenschaub SR, Martini S, Morelli C, Donato F, Volpes R, Pageaux GP, Coilly A, Fagiuoli S, Amaddeo G, Perricone G, Vinaixa C, Berlakovich G, Facchetti R, Polak W, Muiesan P, Duvoux C; European Liver and Intestine Association (ELITA). Delisting of liver transplant candidates with chronic hepatitis C after viral eradication: A European study. J Hepatol. 2016 Sep;65(3):524-31. doi: 10.1016/j.jhep.2016.05.010. Epub 2016 May 17. PMID 27212241
- [Background] Pascasio JM, Vinaixa C, Ferrer MT, Colmenero J, Rubin A, Castells L, Manzano ML, Lorente S, Testillano M, Xiol X, Molina E, Gonzalez-Dieguez L, Oton E, Pascual S, Santos B, Herrero JI, Salcedo M, Montero JL, Sanchez-Antolin G, Narvaez I, Nogueras F, Giraldez A, Prieto M, Forns X, Londono MC. Clinical outcomes of patients undergoing antiviral therapy while awaiting liver transplantation. J Hepatol. 2017 Dec;67(6):1168-1176. doi: 10.1016/j.jhep.2017.08.008. Epub 2017 Aug 24. PMID 28842296
- [Background] Perricone G, Duvoux C, Berenguer M, Cortesi PA, Vinaixa C, Facchetti R, Mazzarelli C, Rockenschaub SR, Martini S, Morelli C, Monico S, Volpes R, Pageaux GP, Fagiuoli S, Belli LS; European Liver and Intestine Transplant Association (ELITA). Delisting HCV-infected liver transplant candidates who improved after viral eradication: Outcome 2 years after delisting. Liver Int. 2018 Dec;38(12):2170-2177. doi: 10.1111/liv.13878. Epub 2018 May 25. PMID 29750389